CLINICAL TRIAL: NCT05808361
Title: Rehabilitation Treatment of Patients With COVID-19 in an Infectious Diseases Hospital, Selection of Patients and Efficacy Criteria: A Retrospective Study With Propensity Score Matching.
Brief Title: Rehabilitation Treatment of Patients With COVID-19
Acronym: COVID-REHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: MEDSI Clinical Hospital 1, ICU (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: COVID-REHAB
Record Dates: First submitted 2023-04-07; First posted 2023-04-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Rehabilitation; Pneumonia, Viral; COVID-19; Quality of Life
MeSH Terms: conditions — Pneumonia, Viral; COVID-19 | interventions — Exercise; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- physical exercise (Experimental): Rehabilitation program includes physical exercises, started in the first 3 days after the patient's body temperature returned to normal.
  Interventions: Other: exercises
- exercises and massage (Experimental): Rehabilitation programs include physical exercises, and chest massage in an electrostatic field, started in the first 3 days after the patient's body temperature returned to normal.
  Interventions: Other: exercises; Other: massage
- Control (No Intervention): Patients received treatment according to the temporary guideline without any rehabilitation program.

INTERVENTIONS:
Other: exercises — The complex of therapeutic exercises included exercises in the initial position lying, sitting and standing. In active and static motor modes under the control of saturation, blood pressure, heart rate and respiratory rate.
  The complex included breathing exercises with the inclusion of compensatory respiratory muscles, elements of sound and drainage gymnastics, and diaphragmatic breathing. Therapeutic gymnastics was carried out in the form of individual lessons with an exercise therapy instructor, a course of 10 procedures, daily, the duration was 20 minutes.
  Arms: exercises and massage; physical exercise
Other: massage — Hardware massage in the electrostatic field with a frequency of 30/60 Hz of the chest area consisted of 10 procedures, daily, the duration of the procedure was 20 minutes.
  Arms: exercises and massage

SUMMARY:
This is single centre retrospective study with propensity score matching. The aim of the study is to develop criteria for determining groups of patients with a new coronavirus infection based on clinical, laboratory and instrumental data for whom rehabilitation programs (physical exercises, chest massage in an electrostatic field) will be effective. Data on predictors of effective rehabilitation in COVID-19 is limited. Knowledge of predictors of possibility and efficacy of rehabilitation programs could enhance patients recovery. The main symptoms of COVID-19 involve the respiratory system and psychological function. Early rehabilitation can reduce hospital length of stay. Different patients have different degrees of dysfunction; therefore, personal plans should be developed according to the patient's age, sex, lifestyle and physical condition. Regular follow-up and rehabilitation guidance were conducted for discharged patients, focusing on improving vital capacity and cardiopulmonary endurance. There is a clear consensus that early rehabilitation is an important strategy for the treatment of polyneuropathy and myopathy in critical disease, to facilitate and improve long-term recovery and patients' functional independence, and to reduce the duration of respiratory support and hospitalization. Early rehabilitation and exercise prescriptions remain to be further optimized, especially for hospitalised patients.

DETAILED DESCRIPTION:
The application of early rehabilitation can promote recovery of body functions; however, further studies are needed to determine the patient selection criteria and relevant mode of rehabilitation program.

A primary concern is regarding the timing of when to start a rehabilitation protocol in the face of the real threat of COVID-19.

Rehabilitation programs include physical exercises, and chest massage in an electrostatic field, started in the first 3 days after the patient's body temperature returned to normal.

The demographic and clinical data will be collected. Laboratory data (white blood cells count, C-reactive protein), and Instrumental data (pulse oxymetry, CT-scan) will be analysed. Rehabilitation evaluation - Health profile according to the quality of life questionnaire before and after each rehabilitation mode will be analysed. Exercise termination criteria: (1) Fluctuations in body temperature > 37.2°C; (2) respiratory symptoms and fatigue worsen; (3) chest tightness, chest pain, breathing difficulties, severe cough, dizziness, headache, blurred vision, palpitations, sweating, trouble standing.

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID-19 admitted to the hospital with mild or moderate COVID-19 (5-50% of lung damage according to CT-scan)

Exclusion Criteria:

* less than 7 days in hospital by any reason,
* chronic decompensated diseases with extrapulmonary organ dysfunction (tumour progression, liver cirrhosis, congestive heart failure), admission to ICU, atonic coma,
* patients in whom more than 30 days have passed since the onset of the disease and before hospitalization,
* patients who received treatment in the intensive care unit, as well as patients who died.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Length of stay in hospital | 30 days
  length of stay in hospital

SECONDARY OUTCOMES:
complete blood count | Change of white blood cells from baseline on day 7 during treatment
  white blood cells
complete blood count dynamics | Change of white blood cells from 7 to 14 day during treatment
  white blood cells
Complaints of fatigue | Change of complains from baseline on day 7 during treatment
  Complaints of fatigue
Complaints of fatigue dynamics | Change of complains from 7 to 14 day during treatment
  Complaints of fatigue
Biochemistry analysis | Change of CRP from baseline on day 7 during treatment
  C-reactive protein (CRP)
Biochemistry analysis dynamics | Change of CRP from 7 to 14 day during treatment
  C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Danil Maliutin, MD, Principal Investigator — Clinical Hospital "MEDSI" in Otradnoe
Locations (1):
- Clinical Hospital "MEDSI" in Otradnoe, Moscow, Russia

REFERENCES:
- [Background] Sun T, Guo L, Tian F, Dai T, Xing X, Zhao J, Li Q. Rehabilitation of patients with COVID-19. Expert Rev Respir Med. 2020 Dec;14(12):1249-1256. doi: 10.1080/17476348.2020.1811687. Epub 2020 Oct 12. PMID 32799694
- [Background] Demeco A, Marotta N, Barletta M, Pino I, Marinaro C, Petraroli A, Moggio L, Ammendolia A. Rehabilitation of patients post-COVID-19 infection: a literature review. J Int Med Res. 2020 Aug;48(8):300060520948382. doi: 10.1177/0300060520948382. PMID 32840156